CLINICAL TRIAL: NCT03331133
Title: Twins Born in Guangzhou Cohort Study
Brief Title: Twins Born in Guangzhou
Acronym: 2-BIG
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Xiu Qiu, Director of the Born in Guangzhou Cohort Study, Guangzhou Women and Children's Medical Center
Other Study IDs: 2017060803
Record Dates: First submitted 2017-10-20; First posted 2017-11-06 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Twin Diseases; Immune Development; Childhood Obesity; Host and Microbiome; Neurodevelopment
Keywords: Twin; Early Development; Cohort
MeSH Terms: conditions — Diseases in Twins; Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During pregnancy: maternal blood, urine and stool At delivery: cord, cord blood and placenta During Infancy：dry blood spot, stool and blood During childhood: blood, buccal swab and stool
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Identical Twins: Twins develop from one zygote with no intervention
  Interventions: Other: No intervention
- Dizygotic Twins: Twins develop from two different zygote with no intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The 2-BIG is a twin birth cohort study located in Guangzhou, China.Its initial aim is to facilitate research on understanding the interplay between genes and environmental factors on disease etiology. Data are collected regarding environmental, family and lifestyle exposures on twins from birth to 18 years old. Biological samples including blood and tissue samples are also collected from the twins and their parents.

DETAILED DESCRIPTION:
Twins share the same intrauterine environment and the early family environment. When conducting research of chronic disease etiology, twins cohort can be a good control of bias from age, gender, genetic and early environment. Twin-based designs provide an estimate of the relative contribution of genetic and non-genetic factors to a specific phenotype. Twins study has an advantage of calculating heritability of traits. Since heritability of traits is various from different populations. It is important to establish database to calculate the heritability of traits associated with chronic major diseases in Chinese population. Twins cohort is rare in China at present. Therefore, extensive information including physical characteristics, mental health, and behaviors is collected from both twins and their parents. Longitudinal follow-up and surveillance of common diseases are also to be conducted. The 2-BIG aims to explore epigenetic markers and genes related to health status, as well as gene-environment interactions on diseases, both in intrauterine and childhood stages, especially in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

1. Live twins delivered in Guangzhou Women and Children's Medical Center
2. Permanent residents or families intended to remain in Guangzhou with their children for no less than 3 years
3. Baseline information during pregnancy available

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Twins delivered in Guangzhou, China and their parents
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopment at early childhood | At age of 1 year old
  Including adaptive, gross motor, fine motor, language, and social function; assessed using Gesell Developmental Schedules.
Intelligence quotient | At age of 6 years old
  Assessed using the Wechsler Preschool and Primary Scale of Intelligence-Fourth Edition including 5 verbal and 3 performance subtests. Intelligence quotient ranges 40-160, in which under 70 is defined as mental retardation. The total score was calculated by an online system.
Change of gene expression during childhood | Age at 1 year , 6 years, 12years and 18years
  DNA methylation, histone acetylation etc. assessed by analyses of blood samples

SECONDARY OUTCOMES:
Change of intestinal flora during early childhood | Age at 6 weeks, 6 months, 1 year , 3 years,6 years, 12years and 18years
  Assessed by analyses of stool samples
Changes of body composition and bone density during early childhood | At birth, age of 6 weeks, 6 months, 1 year , 3 years,6 years, 12years and 18years
  Body composition and bone density are assessed using Dual Energy X-Ray Absorptiometry
Height in kilometer changes during childhood | At birth, age of 6 weeks, 6 months, 1 year, 3 years,6 years, 12years and 18year
  Measured by nurses in clinic
Weight in kilogram changes during childhood | At birth, age of 6 weeks, 6 months, 1 year, 3 years,6 years, 12years and 18year
  Measured by nurses in clinic

CONTACTS AND LOCATIONS:
Overall Officials: Xiu Qiu, PhD, Principal Investigator — Born in Guangzhou Cohort Study in Guangzhou Women and Children's Medical Center
Locations (1):
- Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Qiu X, Lu JH, He JR, Lam KH, Shen SY, Guo Y, Kuang YS, Yuan MY, Qiu L, Chen NN, Lu MS, Li WD, Xing YF, Zhou FJ, Bartington S, Cheng KK, Xia HM. The Born in Guangzhou Cohort Study (BIGCS). Eur J Epidemiol. 2017 Apr;32(4):337-346. doi: 10.1007/s10654-017-0239-x. Epub 2017 Mar 20. PMID 28321694
- See also: Related website — http://www.bigcs.com.cn